CLINICAL TRIAL: NCT01019447
Title: "The Impact of Using Triclosan-antibacterial Sutures on the Incidence of Surgical Site Infection" Prospective, Randomized, Controlled, Double Blind, Multi-centre Study.
Brief Title: The Impact of Using Triclosan-antibacterial Sutures on the Incidence of Surgical Site Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Amygate Healthcare (Unknown)
Responsible Party: Ibrahim Galal Ibrahim, Cairo University Kasr Al-Aini Hospitals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: INDV-0909001
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2009-11

CONDITIONS: Surgical Site Infection
Keywords: Surgical site infection; Antimicrobial triclosan-coated polyglactin 910 suture; Length of hospital stay; SSI
MeSH Terms: conditions — Surgical Wound Infection | interventions — Polyglactin 910

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study group (Active Comparator): The study group in which Triclosan-coated polyglactin 910 antimicrobial sutures will be used.
  Interventions: Other: Vicryl Plus
- Control group (Active Comparator): The control group in which polyglactin 910 antimicrobial sutures will be used.
  Interventions: Other: Vicryl

INTERVENTIONS:
Other: Vicryl Plus — Triclosan-coated polyglactin 910 antimicrobial sutures (Vicryl Plus)
  Other Names: Triclosan-coated polyglactin 910 antimicrobial sutures
  Arms: Study group
Other: Vicryl — Polyglactin 910 antimicrobial sutures (Vicryl)
  Other Names: Polyglactin 910 antimicrobial sutures
  Arms: Control group

SUMMARY:
To compare conventional polyglactin 910 sutures with triclosan-coated polyglactin 910 antimicrobial sutures for the reduction of surgical site infections and any associated health and economic benefits.

ELIGIBILITY:
Inclusion Criteria:

* All patients of different age
* Gender
* Risk factors and procedures candidate for surgical intervention during the period of the study

Exclusion Criteria:

* Patients with an established pre-operative infection at the operative site

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 701 (Actual)
Dates: Start 2009-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Signs of Surgical Site Infections (SSI) according to Centers for Disease Control (CDC) criteria | 30 days (or 1 year in case of prosthesis)

SECONDARY OUTCOMES:
Post-operative hospital stay in days | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Ga Ibrahim, MD, Principal Investigator — Cairo University
Locations (2):
- Egypt (2):
  - Al-Zeraaein Hospital, Cairo, Cairo Governorate
  - Cairo University Kasr Al-Aini Hospital, Cairo, Cairo Governorate